CLINICAL TRIAL: NCT02546505
Title: Impact of Front-of-pack Nutrition Labelling on Consumer Purchases - Controlled Trial in Shopper Laboratory Stores
Brief Title: Impact of Front-of-pack Nutrition Labelling on Consumer Purchases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Paris 13 (Other)
Collaborators: BVA nudge unit (Unknown)
Responsible Party: Principal Investigator, Serge HERCBERG, Professor, University of Paris 13
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: EREN-BVA
Record Dates: First submitted 2015-08-28; First posted 2015-09-11 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Consumer Behavior; Nutrition Labeling
Keywords: Consumer behavior; Nutrition Labeling
MeSH Terms: conditions — Consumer Behavior | interventions — Consumer Health Information

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): The current situation with current way brands show or not nutritional information on Front of Pack (FoP) - without consumer information
- Intervention n°1 (Experimental): Introduction of a Front-of-pack nutrition label (5-CNL) on selected categories of foods. No additional consumer information
  Interventions: Other: Front-of-pack nutrition labeling
- Intervention n°2 (Experimental): Introduction of a Front-of-pack nutrition label (5-CNL) on selected categories of foods. Additional consumer information specifically targeting nutritional information and explaining the 5-CNL will be performed (this information will consist in a concept shown to respondents before the shopping session).
  Interventions: Other: Front-of-pack nutrition labeling; Other: Consumer information

INTERVENTIONS:
Other: Front-of-pack nutrition labeling — Introduction of a Front-of-pack nutrition label (5-CNL) on selected categories of foods.
  Arms: Intervention n°1; Intervention n°2
Other: Consumer information — Information specifically targeting nutritional information and explaining the 5-CNL is presented to the subject (this information will consist in a concept shown to respondents before the shopping session).
  Arms: Intervention n°2

SUMMARY:
Introducing Front-Of-Pack (FOP) nutrition labelling, providing simplified information on nutritional content at a glance, in order to help consumer make informed choices, has been identified as of major interest by public health specialists. In France, a recent report to the Minister of Health has proposed the introduction of a Front-of-Pack nutrition label, the 5-Colour nutrition label. Existing studies on FOP labels mainly focused on assessment of consumers' acceptability/liking and understanding. If most of the studies on purchasing behavior, conducted in real supermarkets, suggested a positive effect of FOP labels on consumers' food choices, the impact of the 5-CNL has not been evaluated.

The main objective is to evaluate the impact of a Front-of-pack nutrition label, the 5-Colour Nutrition Label on consumer purchases in a controlled environment close to real-world settings. Nutritional quality of the items purchased will be compared using the Food Standards Agency nutrient profiling system (FSA score). The study relies on a comparison across three independent samples :

* Control group: The current situation with current way brands show or not nutritional information on Front of Pack (FoP) - without consumer information
* Intervention n°1: Introduction of a Front-of-pack nutrition label (5-CNL) on selected categories of foods. No additional consumer information
* Intervention n°3: Introduction of a Front-of-pack nutrition label (5-CNL) on selected categories of foods. Additional consumer information specifically targeting nutritional information and explaining the 5-CNL will be performed (this information will consist in a concept shown to respondents before the shopping session).

Participants are recruited in the street through quota sampling, based on criteria of gender, age and purchasing habits on the products categories selected for the introduction of the FOP nutrition label.

The study relies on LabStores®, i.e. shopper laboratory stores, which are controlled study spaces in which a store is recreated in reality.The real lab store mimics a store environment with real shelves, product, and cash register, and presents several product categories in a realistic shopping environment. At the end of the shopping session, the respondents proceed to the cashier but don't actually pay for their purchases.

The selected foodstuffs come from actual retailers' brand products available on the French market. Three categories of products were selected, based on expected variability in nutritional quality of the products and logistic criteria (exclusion of fresh products):

* Breakfast cereals
* Sweet biscuits
* Salty snacks The impact of the different labels on nutritional quality (FSA score, calories, lipids, saturated fatty acids, sugars, proteins, fibre, sodium) of the shopping cart is investigated using one way ANOVA. Pairwise comparisons among FOP labels are assessed by using Tukey's multiple comparisons tests.

All tests of significance are two-sided, and a P value <0.05 is considered significant. Statistical analyses are performed using SAS software (version 9.3; SAS Institute Inc.).

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old
* Usually purchasing the selected categories of foods (Breakfast cereals, appetizers, biscuits)

Exclusion Criteria:

* Not used to purchasing the selected categories of foods

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
FSA score to evaluate nutritional quality of the items purchased | Estimated time frame 6 weeks
  Mean Food Standards Agency nutrient profiling system (FSA score) of the items purchased

SECONDARY OUTCOMES:
Energy content of the items purchased | Estimated time frame 6 weeks
  Energy content (Kcal) for 100g of the items purchased
Saturated fatty acid content of the items purchased | Estimated time frame 6 weeks
  Saturated fatty acids content (g) for 100g of the items purchased
Sodium content of the items purchased | Estimated time frame 6 weeks
  Sodium content (mg) for 100g of the items purchased
Sugar content of the items purchased | Estimated time frame 6 weeks
  Sugar content (mg) for 100g of the items purchased
Protein content of the items purchased | Estimated time frame 6 weeks
  Protein content (mg) for 100g of the items purchased
Fiber content of the items purchased | Estimated time frame 6 weeks
  Fiber content (mg) for 100g of the items purchased
Number of purchased items labelled in green/yellow/orange/pink/red | Estimated time frame 6 weeks

REFERENCES:
- [Derived] Julia C, Blanchet O, Mejean C, Peneau S, Ducrot P, Alles B, Fezeu LK, Touvier M, Kesse-Guyot E, Singler E, Hercberg S. Impact of the front-of-pack 5-colour nutrition label (5-CNL) on the nutritional quality of purchases: an experimental study. Int J Behav Nutr Phys Act. 2016 Sep 20;13(1):101. doi: 10.1186/s12966-016-0416-4. PMID 27645372